CLINICAL TRIAL: NCT01637935
Title: Cohort Study of Pioglitazone and Bladder Cancer in Patients With Diabetes
Brief Title: Cohort Study of Pioglitazone and Bladder Cancer in Patients With Type II Diabetes
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Collaborators: Kaiser Permanente (Other); Department of Epidemiology at University of Pennsylvania (Unknown)
Responsible Party: Sponsor
Other Study IDs: 01-03-TL-OPI-524; U1111-1132-3482 (Registry Identifier: WHO)
Record Dates: First submitted 2012-07-07; First posted 2012-07-11 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Diabetes; Bladder Cancer
Keywords: Drug therapy
MeSH Terms: conditions — Diabetes Mellitus; Urinary Bladder Neoplasms | interventions — Pioglitazone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pioglitazone exposed group: Defined as those patients having filled at least two prescriptions for pioglitazone within a 6-month period. Patients in the pioglitazone group may also have exposure to other diabetic medications
  Interventions: Drug: Pioglitazone
- Pioglitazone unexposed group: Defined as patients who did not fill at least two prescriptions for pioglitazone within a 6-month period. Patients in the pioglitazone unexposed group may have been exposed to other diabetic medications. This group also included diabetic patients without any diabetic medications.

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone tablets.
  Other Names: Actos
  Groups: Pioglitazone exposed group

SUMMARY:
To assess the potential association between pioglitazone and bladder cancer compared with non-pioglitazone users among patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Following guidance from the United States Food and Drug Administration (FDA) and European Medicines Agency, the University of Pennsylvania and Kaiser Permanente Northern California (KPNC) designed and conducted this study using the KPNC database to assess the potential association between pioglitazone and bladder cancer among patients with type 2 diabetes mellitus.

The study was conducted over the course of 10 years, with a series of interim analyses undertaken during this period and provided to the sponsor (Takeda) and the appropriate regulatory agencies.

In 2011, the planned 5-year interim analysis of this study was published in Diabetes Care. That report included data from 1 January 1997 to 30 April 2008. Following reporting of these data, there was a request from the FDA for an additional fourth interim analysis at 8 years including data from 1 January 1997 to 31 December 2010.

In August 2011 the FDA requested inclusion of a sensitivity analysis to assess change of cohort entry criteria to minimize left censoring of exposure. Included in the FDA request was a duration analysis for other antidiabetic medications.

In August 2014, the final 10-year analyses were completed and submitted to the sponsor and regulatory agencies.

Interim results previously posted on clinicaltrials.gov are available in the public archive

ELIGIBILITY:
Inclusion Criteria:

* The study cohort included both patients with an established diagnosis of diabetes mellitus prior to January 1, 1997 and those who were newly diagnosed prior to December 31, 2002. Patients were eligible for the study cohort if they met any of the following criteria:

  1. As of January 1, 1997 they had been diagnosed with diabetes mellitus, were age 40 or older and were members of KPNC,
  2. They had been diagnosed with diabetes mellitus, reached age 40 between January 1, 1997 and December 31, 2002 and were KPNC members on their 40th birthday, or
  3. Had diabetes mellitus and were age 40 or older when they joined KPNC between January 1, 1997 and December 31, 2002.

     Exclusion Criteria:
* Diagnosis of bladder cancer recorded in the KPNC cancer registry prior to entry to the cohort or within 6 months of entry into KPNC.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was conducted within Kaiser Permanente Northern California (KPNC), which provides comprehensive healthcare services to approximately 3.2 million members. The source population was identified from the KPNC diabetes registry, which was first constructed in 1993 and has been updated annually since then. The registry identifies patients primarily from four data sources: primary hospital discharge diagnoses of diabetes mellitus (since 1971); two or more outpatient visit diagnoses of diabetes (since 1995); any prescription for a diabetes-related medication (since 1994); or any record of an abnormal hemoglobin A1c (HbA1c) test (>6.7%) (since 1991).
  The diabetes registry gathers data from a variety of KPNC electronic medical records (EMR) to build and follow the registry cohort across time. These data include cancer registries, pharmacy records, laboratory records, and inpatient and outpatient medical diagnoses.
Sampling Method: Probability Sample
Enrollment: 193099 (Actual)
Dates: Start 2004-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

REFERENCES:
- [Result] Lewis JD, Ferrara A, Peng T, Hedderson M, Bilker WB, Quesenberry CP Jr, Vaughn DJ, Nessel L, Selby J, Strom BL. Risk of bladder cancer among diabetic patients treated with pioglitazone: interim report of a longitudinal cohort study. Diabetes Care. 2011 Apr;34(4):916-22. doi: 10.2337/dc10-1068. PMID 21447663
- [Result] Lewis JD, Habel LA, Quesenberry CP, Strom BL, Peng T, Hedderson MM, Ehrlich SF, Mamtani R, Bilker W, Vaughn DJ, Nessel L, Van Den Eeden SK, Ferrara A. Pioglitazone Use and Risk of Bladder Cancer and Other Common Cancers in Persons With Diabetes. JAMA. 2015 Jul 21;314(3):265-77. doi: 10.1001/jama.2015.7996. PMID 26197187
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI
- See also: 10-Year Final Report — https://www.takeda.com/siteassets/en-us/home/external-reference/clinicaltrials.gov/01-03-tl-opi-524-10-year_final_report.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Not applicable (database study)
Pre-assignment Details: Not applicable (database study)
Groups:
- Pioglitazone Exposed Group: Patients ever exposed to pioglitazone.
- Pioglitazone Unexposed Group: Patients never exposed to pioglitazone.
Period: Overall Study
Arm/Group | Pioglitazone Exposed Group | Pioglitazone Unexposed Group
Started | 34181 | 158918
Completed | 34181 | 158918
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone Exposed Group | Pioglitazone Unexposed Group | Total
Number analyzed (Participants) | 34181 | 158918 | 193099
Age, Customized [Number; unit: percentage of participants]
  40-49 years | 29.2 | 22.1 | 51.3
  50-59 years | 33.0 | 25.6 | 58.6
  60-69 years | 25.7 | 26.2 | 51.9
  70 years and older | 12.0 | 26.1 | 38.1
Sex/Gender, Customized [Number; unit: percentage of participants]
  Female | 46.5 | 46.5 | 93
  Male | 53.5 | 53.5 | 107
Race/Ethnicity, Customized [Number; unit: percentage of participants]
  White | 51.3 | 52.3 | 103.6
  Black | 10.2 | 10.8 | 21
  Asian | 14.8 | 12.8 | 27.6
  Hispanic | 13.4 | 10.6 | 24
  Other | 5.9 | 5.7 | 11.6
  Missing | 4.3 | 7.8 | 12.1
Current smoker [Number; unit: percentage of participants] | 20.4 | 17.4 | 37.8
Renal function at baseline [Number; unit: percentage of participants] — Elevated creatinine: Creatinine >1.4 mg/dL for women and >1.5 mg/dL for men.
  percentage of participants
    Normal creatinine | 77.4 | 77.1 | 154.5
    Elevated creatinine | 4.0 | 8.7 | 12.7
    Missing | 18.6 | 14.1 | 32.7
Congestive heart failure at baseline [Number; unit: percentage of participants] | 3.0 | 6.9 | 9.9
Baseline Glycosylated Hemoglobin (HbA1c) [Number; unit: percentage of participants]
  <7% | 17.1 | 28.6 | 45.7
  7-7.9% | 18.3 | 19.3 | 37.6
  8-8.9% | 12.8 | 10.4 | 23.2
  9-9.9% | 9.7 | 7.0 | 16.7
  ≥10% | 23.9 | 17.1 | 41
  Missing | 18.1 | 17.5 | 35.6
Newly diagnosed with diabetes mellitus at the start of follow-up [Number; unit: percentage of participants] — Includes newly diagnosed patients and patients who newly enrolled in Kaiser Permanente with an existing diagnosis of diabetes mellitus.
  percentage of participants | 50.8 | 57.9 | 108.7
Diabetes duration at baseline [Number; unit: percentage of participants]
  0-4 years | 60.1 | 62.8 | 122.9
  5-9 years | 9.2 | 6.0 | 15.2
  10 or more years | 9.1 | 10.9 | 20
  Missing | 21.6 | 20.4 | 42
Other cancer prior to baseline [Number; unit: percentage of participants] | 3.1 | 5.3 | 8.4
Other diabetes medications [Number; unit: percentage of participants] — Includes use of any other diabetes medications during follow-up.
  percentage of participants
    Other thiazolidinediones | 8.2 | 1.5 | 9.7
    Metformin | 84.8 | 45.9 | 130.7
    Sulfonylureas | 89.8 | 61.2 | 151
    Other oral hypoglycemic drugs | 6.4 | 1.4 | 7.8
    Insulin | 52.7 | 29.4 | 82.1
    Never treated with any diabetes medication | 0.0 | 14.3 | 14.3

OUTCOME MEASURES:

1. Primary Outcome: Incident Diagnosis of Bladder Cancer (10-year Analysis)
Description: Incident bladder cancers were identified from January 1, 1997 to December 31, 2012.
Time Frame: January 1, 1997 to December 31, 2012
Population: All participants.
Measure: Number (95% Confidence Interval); unit: events per 100,000 person years
Arm/Group | Pioglitazone Exposed Group | Pioglitazone Unexposed Group
Number analyzed (Participants) | 34181 | 158918
events per 100,000 person years | 89.8 [76.9 to 102.7] | 75.9 [71.3 to 80.4]
Statistical Analysis 1: Comparison: Pioglitazone Exposed Group vs Pioglitazone Unexposed Group; Fully adjusted refers to inclusion of all potential confounders in the statistical model from the 5-year interim report plus year of cohort entry: age, sex, race/ethnicity, other diabetes medications, smoking, other bladder conditions, median household income, congestive heart failure, cancer other than bladder cancer, renal insufficiency, HbA1c and the interaction with new diagnosis of diabetes, duration of diabetes, and year of cohort entry; Test type: Superiority or Other; Cox Proportional Hazard = 1.10, 95% CI [0.92 to 1.31]
Statistical Analysis 2: Comparison: Pioglitazone Exposed Group vs Pioglitazone Unexposed Group; Fully adjusted adding the proteinuria testing variable; Test type: Superiority or Other; Cox Proportional Hazard = 1.06, 95% CI [0.89 to 1.26]

2. Secondary Outcome: Incident Diagnosis of Bladder Cancer by Time Since Starting Pioglitazone (10 Year Analysis)
Time Frame: January 1, 1997 to December 31, 2012
Measure: Number (95% Confidence Interval); unit: events per 100,000 person years
Arm/Group | Pioglitazone Exposed Group | Pioglitazone Unexposed Group
Number analyzed (Participants) | 34181 | 158918
events per 100,000 person years
  Less than 4.5 years | 68.2 [54.0 to 82.5] | NA [NA to NA] — Not calculated for the No Pioglitazone Treatment group.
  4.5 -8.5 years | 111.6 [84.5 to 138.7] | NA [NA to NA] — Not calculated for the No Pioglitazone Treatment group.
  More than 8.0 years | 125.8 [82.9 to 168.7] | NA [NA to NA] — Not calculated for the No Pioglitazone Treatment group.
Statistical Analysis 1: Comparison: Pioglitazone Exposed Group vs Pioglitazone Unexposed Group; Time since starting pioglitazone <4.5 years vs unexposed group. Fully adjusted including all potential confounders in statistical model from 5-year interim report plus year of cohort entry: age, sex, race/ethnicity, other diabetes medications, smoking, other bladder conditions, median household income, congestive heart failure, cancer other than bladder, renal insufficiency, HbA1c and interaction with new diagnosis of diabetes, duration of diabetes, year of cohort entry and proteinuria; Test type: Superiority or Other; Hazard Ratio (HR) = 0.89, 95% CI [0.71 to 1.12]
Statistical Analysis 2: Comparison: Pioglitazone Exposed Group vs Pioglitazone Unexposed Group; Time since starting pioglitazone 4.5-8 years vs unexposed group. Fully adjusted including all potential confounders in statistical model from 5-year interim report plus year of cohort entry: age, sex, race/ethnicity, other diabetes medications, smoking, other bladder conditions, median household income, congestive heart failure, cancer other than bladder, renal insufficiency, HbA1c and interaction with new diagnosis of diabetes, duration of diabetes, year of cohort entry and proteinuria; Test type: Superiority or Other; Hazard Ratio (HR) = 1.21, 95% CI [0.93 to 1.59]
Statistical Analysis 3: Comparison: Pioglitazone Exposed Group vs Pioglitazone Unexposed Group; Time since starting pioglitazone >8 years vs unexposed group. Fully adjusted including all potential confounders in statistical model from 5-year interim report plus year of cohort entry: age, sex, race/ethnicity, other diabetes medications, smoking, other bladder conditions, median household income, congestive heart failure, cancer other than bladder, renal insufficiency, HbA1c and interaction with new diagnosis of diabetes, duration of diabetes, year of cohort entry and proteinuria; Test type: Superiority or Other; Hazard Ratio (HR) = 1.20, 95% CI [0.83 to 1.75]

3. Secondary Outcome: Incident Diagnosis of Bladder Cancer by Duration of Pioglitazone Therapy (10 Year Analysis)
Time Frame: January 1, 1997 to December 31, 2012
Population: All participants.
Measure: Number (95% Confidence Interval); unit: events per 100,000 person years
Arm/Group | Pioglitazone Exposed Group | Pioglitazone Unexposed Group
Number analyzed (Participants) | 34181 | 158918
events per 100,000 person years
  Less than 1.5 years | 67.5 [50.4 to 84.6] | NA [NA to NA] — Not calculated for the No Pioglitazone Treatment group.
  1.5 - 4.0 years | 88.4 [67.5 to 109.3] | NA [NA to NA] — Not calculated for the No Pioglitazone Treatment group.
  More than 4 years | 113.7 [84.2 to 143.2] | NA [NA to NA] — Not calculated for the No Pioglitazone Treatment group.
Statistical Analysis 1: Comparison: Pioglitazone Exposed Group vs Pioglitazone Unexposed Group; Duration of therapy <1.5 years. Fully adjusted including all potential confounders in statistical model from 5-year interim report plus year of cohort entry: age, sex, race/ethnicity, other diabetes medications, smoking, other bladder conditions, median household income, congestive heart failure, cancer other than bladder, renal insufficiency, HbA1c and interaction with new diagnosis of diabetes, duration of diabetes, year of cohort entry and proteinuria; Test type: Superiority or Other; Hazard Ratio (HR) = 0.88, 95% CI [0.68 to 1.16]
Statistical Analysis 2: Comparison: Pioglitazone Exposed Group vs Pioglitazone Unexposed Group; Duration of therapy 1.5-4 years. Fully adjusted including all potential confounders in statistical model from 5-year interim report plus year of cohort entry: age, sex, race/ethnicity, other diabetes medications, smoking, other bladder conditions, median household income, congestive heart failure, cancer other than bladder, renal insufficiency, HbA1c and interaction with new diagnosis of diabetes, duration of diabetes, year of cohort entry and proteinuria; Test type: Superiority or Other; Hazard Ratio (HR) = 1.03, 95% CI [0.80 to 1.33]
Statistical Analysis 3: Comparison: Pioglitazone Exposed Group vs Pioglitazone Unexposed Group; Duration of therapy >4 years. Fully adjusted including all potential confounders in statistical model from 5-year interim report plus year of cohort entry: age, sex, race/ethnicity, other diabetes medications, smoking, other bladder conditions, median household income, congestive heart failure, cancer other than bladder, renal insufficiency, HbA1c and interaction with new diagnosis of diabetes, duration of diabetes, year of cohort entry and proteinuria; Test type: Superiority or Other; Hazard Ratio (HR) = 1.16, 95% CI [0.87 to 1.54]

4. Secondary Outcome: Incident Diagnosis of Bladder Cancer by Cumulative Dose of Pioglitazone (10 Year Analysis)
Time Frame: January 1, 1997 to December 31, 2012
Population: All participants.
Measure: Number (95% Confidence Interval); unit: events per 100,000 person years
Arm/Group | Pioglitazone Exposed Group | Pioglitazone Unexposed Group
Number analyzed (Participants) | 34181 | 158918
events per 100,000 person years
  1 - 14000 mg | 69.1 [52.4 to 85.8] | NA [NA to NA] — Not calculated for the No Pioglitazone Treatment group.
  14001 - 40000 mg | 96.9 [74.0 to 119.8] | NA [NA to NA] — Not calculated for the No Pioglitazone Treatment group.
  >40000 mg | 101.4 [73.5 to 129.2] | NA [NA to NA] — Not calculated for the No Pioglitazone Treatment group.
Statistical Analysis 1: Comparison: Pioglitazone Exposed Group vs Pioglitazone Unexposed Group; Cumulative dose 1-14000 mg. Fully adjusted including all potential confounders in statistical model from 5-year interim report plus year of cohort entry: age, sex, race/ethnicity, other diabetes medications, smoking, other bladder conditions, median household income, congestive heart failure, cancer other than bladder, renal insufficiency, HbA1c and interaction with new diagnosis of diabetes, duration of diabetes, year of cohort entry and proteinuria; Test type: Superiority or Other; Hazard Ratio (HR) = 0.90, 95% CI [0.69 to 1.16]
Statistical Analysis 2: Comparison: Pioglitazone Exposed Group vs Pioglitazone Unexposed Group; Cumulative dose 14001-40000 mg. Fully adjusted including all potential confounders in statistical model from 5-year interim report plus year of cohort entry: age, sex, race/ethnicity, other diabetes medications, smoking, other bladder conditions, median household income, congestive heart failure, cancer other than bladder, renal insufficiency, HbA1c and interaction with new diagnosis of diabetes, duration of diabetes, year of cohort entry and proteinuria; Test type: Superiority or Other; Hazard Ratio (HR) = 1.10, 95% CI [0.85 to 1.42]
Statistical Analysis 3: Comparison: Pioglitazone Exposed Group vs Pioglitazone Unexposed Group; Cumulative dose >40000 mg. Fully adjusted including all potential confounders in statistical model from 5-year interim report plus year of cohort entry: age, sex, race/ethnicity, other diabetes medications, smoking, other bladder conditions, median household income, congestive heart failure, cancer other than bladder, renal insufficiency, HbA1c and interaction with new diagnosis of diabetes, duration of diabetes, year of cohort entry and proteinuria; Test type: Superiority or Other; Hazard Ratio (HR) = 1.07, 95% CI [0.79 to 1.44]

5. Secondary Outcome: Stage of Bladder Cancer (10 Year Analysis)
Time Frame: January 1, 1997 to December 31, 2012
Population: Participants diagnosed with bladder cancer.
Measure: Number; unit: percentage of participants
Arm/Group | Pioglitazone Exposed Group | Pioglitazone Unexposed Group
Number analyzed (Participants) | 186 | 1075
percentage of participants
  PUNLMP | 1 | 1
  In situ | 50 | 49
  Local | 40 | 38
  Regional | 4 | 6
  Distant | 2 | 3
  Undetermined | 3 | 3

ADVERSE EVENTS:
Description: Adverse events not applicable as this study is based on the secondary use of electronic medical records.
Arm/Group | Pioglitazone Exposed Group | Pioglitazone Unexposed Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 45 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.